CLINICAL TRIAL: NCT00315406
Title: Longitudinal Protocol of Polyarteritis Nodosa
Brief Title: Determining Disease Activity Biomarkers in Individuals With Polyarteritis Nodosa
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Principal Investigator, Peter Merkel, Professor, University of Pennsylvania
Other Study IDs: VCRC5504; U54AR057319 (NIH)
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Polyarteritis Nodosa
Keywords: PAN; Periarteritis Nodosa
MeSH Terms: conditions — Polyarteritis Nodosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum and plasma), urine, and DNA
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Polyarteritis nodosa (PAN) is a rare immune system disorder that causes swelling and damage to small- and medium-sized blood vessels in the body. In order to properly treat this disease, it is critical that the level of disease activity can be determined over the course of the disease. The purpose of this study is to determine new biological markers, or biomarkers, that may be used to assess the severity of disease in people with PAN.

DETAILED DESCRIPTION:
PAN, also known as systemic necrotic vasculitis, was the first recognized form of primary systemic vasculitis. PAN causes the inflammation of small- to medium-sized blood vessels, especially those supplying the nerves, skin, kidneys, gastrointestinal tract, heart, eye, and genitals. Unlike another form of vasculitis called microscopic polyangiitis, PAN does not usually cause glomerulonephritis, a type of kidney disease, or vasculitis in the very smallest blood vessels (arterioles, capillaries, and venules). There are no radiographic or serologic tests that can reliably measure disease activity in PAN. Currently, clinicians must rely on patients' symptoms, signs, laboratory tests, and imaging to guide treatment decisions, but such data are rarely consistently reliable in determining PAN disease activity. This study will use new scientific methods to discover new biomarkers that can be used to monitor disease activity in PAN patients. These biomarkers may be used to help direct clinical care for PAN patients and assist in future drug development.

Study visits will occur monthly for the first year, then every 3 months thereafter for the remainder of the study. Blood and urine collection will occur at every visit. A physical exam and medical and medication history will occur every 3 months; also, participants will be asked to complete several questionnaires to assess disease activity, health status, and tobacco, alcohol, and drug use. Participants may have additional study visits if a disease flare or disease-related complications occur during the study.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian willing to provide informed consent, if applicable
* Diagnosis of vasculitis
* Diagnosis of PAN, meeting at least 1 major criterion and 1 minor criterion OR 2 major criteria of the following adapted American College of Rheumatology (ACR) criteria that fall under the diagnosis of PAN and that are not explained by other causes:

MAJOR CRITERIA

1. Arteriographic abnormality
2. Presence of granulocyte or mixed leukocyte infiltrate in an arterial wall on biopsy
3. Mononeuropathy or polyneuropathy

MINOR CRITERIA

1. Weight loss of more than 4 kg (8.8 lbs)
2. Livedo reticularis, cutaneous ulcerations, or skin nodules
3. Testicular pain or tenderness
4. Myalgias
5. Diastolic blood pressure greater than 90 mm Hg
6. Elevated blood urea nitrogen (BUN) or serum creatinine levels
7. Ischemic abdominal pain

Exclusion Criteria:

* Microscopic polyangiitis
* Granulomatosis with polyangiitis(Wegener's)
* Eosinophilic granulomatosis with polyangiitis (Churg-Strauss)
* Takayasu's arteritis
* Giant cell arteritis
* Cogan's syndrome
* Behcet's disease
* Sarcoidosis
* Kawasaki disease
* Cryoglobulinemic vasculitis
* Systemic lupus erythematosus
* Rheumatoid arthritis
* Mixed connective tissue disease or any overlap autoimmune syndrome
* Presence of antiproteinase 3 or antimyeloperoxidase antineutrophil cytoplasmic antibodies (ANCA)
* Glomeronephritis
* Alveolar hemorrhage
* Hepatitis B, hepatitis C, or HIV infection
* Any other infectious form of medium vessel vasculitis
* Isolated cutaneous PAN

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with polyarteritis nodosa. Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2006-04 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Discover biomarkers in PAN capable of measuring disease activity and response to treatment. | Study completion

SECONDARY OUTCOMES:
Measure the predictive value of biomarkers for clinical outcome in PAN. | Study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter A. Merkel, MD, MPH, Study Chair — University of Pennsylvania
Locations (9):
- United States (7):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University School of Medicine, Boston, Massachusetts
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonsib SM. Polyarteritis nodosa. Semin Diagn Pathol. 2001 Feb;18(1):14-23. PMID 11296989
- [Background] Said G, Lacroix C. Primary and secondary vasculitic neuropathy. J Neurol. 2005 Jun;252(6):633-41. doi: 10.1007/s00415-005-0833-9. Epub 2005 Apr 5. PMID 15806339
- See also: Vasculitis Clinical Research Consortium — http://rarediseasesnetwork.org/cms/vcrc/
- See also: Rare Diseases Clinical Research Network — http://rarediseasesnetwork.org/